CLINICAL TRIAL: NCT03788421
Title: Comparison Between 2 Techniques for Bilateral Salpingectomy During Cesarean Section
Brief Title: Comparison Between 2 Techniques for Bilateral Salpingectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yaniv Zipori MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0427 - 18 - RMB
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Sterility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Constriction; Sutures

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Women undergoing elective bilateral salpingectomy during cesarean section with LIGASURE.
  Interventions: Device: LIGASURE
- Control group (Active Comparator): Women undergoing elective bilateral salpingectomy during cesarean section with traditional step by step clamping and suturing.
  Interventions: Procedure: Clamping and suturing

INTERVENTIONS:
Device: LIGASURE — Electricity based cautery tool used during both laparoscopic and open surgery for optimal hemostasis.
  Arms: Study group
Procedure: Clamping and suturing — Step by step clamping and suturing of the mesosalpinx until achievement of total salpingectomy.
  Arms: Control group

SUMMARY:
A comparison between 2 techniques for bilateral salpingectomy during cesarean section.

Primary outcomes are total operative time and bilateral completion of the randomized procedure. Secondary outcomes included surgical complications and post operation complications.

DETAILED DESCRIPTION:
Ovarian cancer is the most lethal gynecologic malignancy. Major contributors to this high mortality are the lack of effective screening strategies, diagnosis at advanced stage of presentation as well as the high risk of recurrence. In the last years the Gynecologic Associations worldwide have recommended that total salpingectomy be considered for potential ovarian cancer risk reduction in benign gynecologic surgeries after completion of childbearing.

However, the data are limit regarding the Preferred surgical technique during cesarean section.

In this randomized controled trial the investigators will compare between various techniques for bilateral salpingectomy during cesarean section.

Primary outcomes are total operative time and bilateral completion of the randomized procedure. Secondary outcomes included surgical complications and post operation complications.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing elective Cesarean Section and are interested and have signed informed consent regarding bilateral salpingectomy.

Exclusion Criteria:

* Inability to give informed consent.
* Preterm delivery (< 37 weeks' gestation).
* Fetal demise.
* Prenatal diagnosis of fetal or placental abnormalities.
* Previous tubal surgery.
* The use of anticoagulants.
* Associated immunosuppressive conditions.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 51 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Total salpingectomy time. | Up to 1 week from recruitment
  Time in minutes from beginning of salpingectomy procedure until end of the salpingectomy procedure.

SECONDARY OUTCOMES:
Bleeding during salpingectomy | Up to 4 hours from the beginning of the procedure
  Estimated amount of bleeding in milliliters during the salpingectomy procedure
Bleeding during cesarean section | Up to 4 hours from the beginning of the procedure
  Estimated amount of bleeding in milliliters during the whole cesarean section.
Hemoglobin level | Up to 5 days from surgery
  Changes in hemoglobin level before and after surgery
Blood transfusion rate | Up to 5 days from surgery
  The rate of blood transfusion post cesarean section
Postoperative stay | Up to 2 weeks from surgery
  The length of maternal postoperative stay.
Visual analogue score | Up to 2 weeks from surgery
  Pain scoring between 0-10 post-surgery
Wound complications | Up to 2 weeks from surgery
  The rate of wound complications postpartum.
Need for opioids | Up to 2 weeks from surgery
  The rate of opioid treatment postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Zipori, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No